CLINICAL TRIAL: NCT03973320
Title: Outcomes After Hypotensive Neuraxial Anesthesia in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-2235
Record Dates: First submitted 2019-05-28; First posted 2019-06-04 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-03

CONDITIONS: Total Hip Arthroplasty; Primary Total Hip Arthroplasty; Hypotension; Database
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Total Hip Arthroplasty: This is a chart review to determine if hypotensive neuraxial anesthesia is associated with worse outcomes in Primary Total Hip Arthroplasty
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — This is a chart review to determine if hypotensive neuraxial anesthesia is associated with worse outcomes in Primary Total Hip Arthroplasty patients.

SUMMARY:
This is a retrospective chart review to determine if neuraxial anesthesia is associated with worse outcomes after Primary Total Hip Arthroplasty.

DETAILED DESCRIPTION:
The goal of this study is to determine if hypotensive neuraxial anesthesia is associated with worse outcomes in Primary Total Hip Arthroplasty. The plan to analyze the outcomes is listed below:

Primary outcomes:

Multiple logistic regression will be used to compute the adjusted odds ratios of any postoperative complications (MI, CVA, death) , adjusting for covariates including duration of intraoperative mean arterial pressure of less than pre-defined threshold, such as 55, or 60 mmHg mean blood pressure.

Sensitivity analyses will also consider the effects of intra-operative hypotension (IOH) defined as mean blood pressure of less than 40, 45, 50, 55, 60, and 65 mm Hg.

Secondary outcomes:

Multiple logistic regression will be to compute the adjusted odds ratios of individual postoperative complications, (such as MI, CVA, stroke) , adjusting for covariates including duration of intraoperative mean blood pressure of less than pre-defined threshold, such as 55, or 60 mmHg mean blood pressure. Sensitivity analyses will also be conducted to test the effects of extend of IOH on complications.

ELIGIBILITY:
Inclusion Criteria:

* All primary total hip arthroplasty patient data with sufficiently complete intraoperative vital signs

Exclusion Criteria:

* Revision primary total hip arthroplasty
* Incomplete intraoperative vital signs
* Anterior total hip arthroplasty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Primary Total Hip Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 11292 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiabin Liu, MD, PhD, Principal Investigator — Hospital for Special Surgey
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Total Hip Arthroplasty
Started | 11292
Completed | 11292
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Primary Total Hip Arthroplasty Without Complications; Primary Total Hip Arthroplasty With Common Complications: This is a chart review to determine if hypotensive neuraxial anesthesia is associated with worse outcomes in Primary Total Hip Arthroplasty
  Chart Review: This is a chart review to determine if hypotensive neuraxial anesthesia is associated with worse outcomes in Primary Total Hip Arthroplasty patients.
- Total: Total of all reporting groups
Arm/Group | Primary Total Hip Arthroplasty Without Complications | Primary Total Hip Arthroplasty With Common Complications | Total
Number analyzed (Participants) | 11224 | 68 | 11292
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 71.5] | 75.6 [63.1 to 81.6] | 64 [57 to 71.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5955 | 30 | 5985
  Male | 5269 | 38 | 5307
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 9842 | 49 | 9891
BMI (Body Mass Index) [Median (Inter-Quartile Range); unit: kg/m^2] | 28.1 [24.8 to 32.1] | 28 [25.1 to 33.3] | 28.1 [24.8 to 32.2]
Anesthetic type: Spinal [Count of Participants; unit: Participants] | 3584 | 16 | 3600
Anesthetic type: Epidural/CSE [Count of Participants; unit: Participants] | 7640 | 52 | 7692
ASA of 1 & 2 [Count of Participants; unit: Participants] — The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities.
  ASA I A normal healthy patient. ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life.
  Patients are given an ASA prior to surgery and this is listed on their EPIC chart.
  Participants | 9254 | 37 | 9291
ASA of 3 [Count of Participants; unit: Participants] | 1970 | 31 | 2001

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Myocardial Infarction, Cerebrovascular Accident, or Mortality
Description: The association between levels and length of intraoperative controlled hypotension and incidence rates of individual and composite outcome of any of the following events: (i) myocardial infarction (MI), (ii) cerebrovascular accident (CVA), (iii) death. If any of these events are positive, then the composite outcome will be positive. The units of measurement will be the same.
Time Frame: Day of Surgery (Day 0) through discharge (days til discharge is an average of 2 days), follow-ups up to 30 days post-surgery
Population: 21 patients out of 11,292 fit complication definition.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Total Hip Arthroplasty
Number analyzed (Participants) | 21
Participants
  Myocardial Infarction | 16
  Stroke | 2
  In-Hospital mortality | 0
  30-day mortality | 3

ADVERSE EVENTS:
Time Frame: The time period to which adverse events (i.e. deaths) were collected was up to 30 days following a total hip arthroplasty surgery.
Description: The primary outcome was "the incidences of (i) myocardial infarction (MI), (ii) cerebrovascular accident (CVA), (iii) death, and (iv) calculated perioperative intraoperative blood loss", and these events were recorded retrospectively. As a result, none of the three types of adverse events posed a risk to participants. This study collects past information and no new data was actively collected from individuals.
Arm/Group | Primary Total Hip Arthroplasty
All-Cause Mortality (participants affected / at risk) | 3/11292
Serious Adverse Events (participants affected / at risk) | 0/11292
Other Adverse Events (participants affected / at risk) | 18/11292
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Total Hip Arthroplasty (N=11292)
Myocardial Infarction (Cardiac disorders) | 16
Stroke (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03973320/Prot_SAP_000.pdf